CLINICAL TRIAL: NCT06215352
Title: Influence of Chrono-nutrition Factors, Temporal Dietary Patterns, and Their Interactions With Dietary Quality During Pregnancy on Maternal Gestational Diabetes, Glycemic Parameters, and Gestational Weight Gain.
Brief Title: Influence of Chrono-nutrition Factors and Temporal Dietary Patterns on Glycemic Parameters During Pregnancy.
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202301101RIND
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Chrono-nutrition; Gestational diabetes mellitus; Metabolic health
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will first freeze the blood samples for future analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Chrono-nutrition factors — Dietary records would be used to assess the chrono-nutrition factors such as night eating, breakfast skipping, meal frequency, and daily fasting.

SUMMARY:
This study aims to establish a new cohort study to investigate the relationship between chrono-nutrition factors during pregnancy and maternal GDM (Gestational diabetes mellitus), glycemic parameters, and gestational weight gain.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM), characterized by hyperglycemia first diagnosed during pregnancy, is associated with an increased risk of full-fledged type 2 diabetes (T2D) in mothers and adverse metabolic health in their offspring. In Taiwan, the prevalence of GDM has risen from 7.6% in 2004 to 13.4% in 2015, affecting approximately 1 in 7 pregnancies. Even at levels below the diagnostic threshold for GDM, studies such as the Hyperglycemia and Adverse Pregnancy Outcomes (HAPO) have shown a clear graded relationship between higher maternal glycemia and an elevated risk of adverse birth outcomes and childhood insulin resistance.

Metabolic health and glycemic profile of mothers are in turn heavily influenced by diet and nutrition. While dietary content is crucial, multiple lines of evidence now suggests that not only what one eats but also when one eats impacts health. The master circadian clock in the human brain orchestrates circadian rhythms in response to the light-dark cycle. However, it is now recognized that most organs possess peripheral circadian clocks that are strongly influenced by behavioral rhythms, including feeding/fasting, activity/rest, and wake/sleep cycles. Chrono-nutrition is an emerging field of study concerning the interplay between the endogenous circadian rhythm, dietary intake, metabolism, and health. There are various dimensions of chrono-nutrition including meal timing, frequency, and regularity, and daily fasting duration. These individual dimensions have been linked to health outcomes, but few studies have examined the intricate interconnectedness across these different dimensions. Another research gap is that there is a dearth of studies investigating chrono-nutrition factors in pregnant populations.

Thus, to address these research gaps, the investigators aim to establish a new cohort study to investigate the relationship between chrono-nutrition factors during pregnancy and maternal GDM, glycemic parameters, and gestational weight gain.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 20 years or older.
2. Pregnancy duration between 10 and 15 weeks.

Exclusion Criteria:

1. Diagnosis of type 1 diabetes, type 2 diabetes, or gestational diabetes.
2. Currently taking medications that may affect glucose metabolism (e.g., metformin).
3. Irregular working schedule, such as shift work.
4. Presence of a multiple pregnancy.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women attending first antenatal clinic visits at National Taiwan University Hospital (NTUH) will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 316 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Glycemic Parameters | 2 hours
  Values derived from oral glucose tolerance test (OGTT), including fasting, 1-hour, and 2-hour glucose levels, and gestational diabetes diagnosis.
Gestational weight gain | 1 minutes
  Institute of Medicine guideline will be applied to classify gestational weight gain adequacy based on pre-pregnancy body mass index categories.

CONTACTS AND LOCATIONS:
Overall Officials: Ling-Wei Chen, Ph.D., Principal Investigator — Institute of Epidemiology and Preventive Medicine, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng District, Taiwan